CLINICAL TRIAL: NCT00982735
Title: An Observational Cohort Study to Evaluate the Safety and Efficacy of Micardis Tablets Taken Once Daily at 40 mg/Day and 80 mg/Day in Hypertensive Patients Under Real Life Conditions in Usual Clinical Practice.
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 502.540
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2010-03-24 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The "CONTROL" study is an out patient based prospective observational cohort study. The main aim of the study is to survey the safety and efficacy of Micardis 40 mg/day and 80 mg/day under real life conditions in usual clinical practice in essential hypertensive patients in the Kingdom of Saudi Arabia. The patients participating in the study will be surveyed for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Aged 20 to 80 years old.
* Adult essential hypertensive either newly diagnosed and untreated, or previously treated and uncontrolled patients; sitting blood pressure: systolic BP > 140 mmHg but < 180 mmHg, and/or diastolic BP > 90 mmHg but < 110 mmHg).
* Patients who are assessed to benefit from the intake of angiotensin II receptor blocker (ARB) monotherapy or as add-on medication.

Exclusion Criteria:

* Patients with contraindications to telmisartan use (as per the Micardis® Tablets package insert).
* Known hypersensitivity to the active ingredient or to any of the excipients of Micardis® Tablets.
* Any other clinical condition which, in the opinion of the attending physician, would not allow safe administration of the study medications.
* Patients participating in any other protocol

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Essential hypertensive patients
Sampling Method: Non-Probability Sample
Enrollment: 987 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Groups:
- Telmisartan 40mg or Telmisartan 80 mg Once a Day: Telmisartan (Micardis) 40mg (Telmisartan (Micardis) 80 mg) once a day
Period: Overall Study
Arm/Group | Telmisartan 40mg or Telmisartan 80 mg Once a Day
Started | 987
Completed | 757
Not Completed | 230
Not completed — Lost to Follow-up | 6
Not completed — Patient ineligible for trial | 224

BASELINE CHARACTERISTICS:
Arm/Group | Telmisartan 40mg or Telmisartan 80 mg Once a Day
Number analyzed (Participants) | 987
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.12 (8.54)
Gender [Number; unit: participants] — Data with regards to gender is not available for 27 out of the total number of 987 participants.
  participants
    Female | 313
    Male | 647

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Blood Pressure (BP) Control, Sitting Diastolic BP Over Systolic BP 90 Over 140 mm Hg and/or Reduction From Baseline in Sitting Systolic BP or Diastolic BP More Than 10 mm Hg.
Time Frame: 24 weeks
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40mg or Telmisartan 80 mg Once a Day
Number analyzed (Participants) | 757
Participants | 711

2. Secondary Outcome: Assessment by Attending Physicians on the Effectiveness of Treatment With Telmisartan, According to Their Opinion
Description: A 5-point scale was used by the attending physicians to assess the effectiveness of Telmisartan according to their opinion. The scale was rated from 0 (not satisfactory), 1 (marginal), 2 (satisfactory), 3 (very satisfactory) to 4 (outstanding).
Time Frame: 24 weeks
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40mg or Telmisartan 80 mg Once a Day
Number analyzed (Participants) | 757
Participants
  Marginal | 21
  Not satisfactory | 3
  Outstanding | 221
  Satisfactory | 159
  Very satisfactory | 363

3. Secondary Outcome: Change From Baseline in Microalbuminuria at 24 Weeks
Time Frame: Baseline and 24 weeks
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40mg or Telmisartan 80 mg Once a Day
Number analyzed (Participants) | 757
Participants
  No microalbuminuria at baseline (BL) and at week24 | 433
  No microalbuminuria BL and 30 mg/g Crea at week24 | 5
  No microalbuminuria BL and 100 mg/g Crea at week24 | 1
  No microalbuminuria BL and 500 mg/g Crea at week24 | 0
  30 mg/g Crea BL and no microalbuminuria at week24 | 111
  30mg/g Crea at BL and at week24 | 25
  30mg/g Crea at BL and 100mg/g Crea at week24 | 1
  30mg/g Crea at BL and 500mg/g Crea at week24 | 0
  100 mg/g Crea BL and no microalbum.uria at week24 | 58
  100mg/g Crea at BL and 30mg/g Crea at week24 | 84
  100mg/g Crea at BL and at week24 | 11
  100mg/g Crea at BL and 500mg/g Crea at week24 | 0
  500mg/g Crea at BL + no microalbuminuria at week24 | 8
  500mg/g Crea at BL + 30mg/g Crea at week24 | 7
  500mg/g Crea at BL and 100mg/g Crea at week24 | 12
  500mg/g Crea at BL and at week24 | 1

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Telmisartan 40mg or Telmisartan 80 mg Once a Day
Serious Adverse Events (participants affected / at risk) | 0/757
Other Adverse Events (participants affected / at risk) | 0/757

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.